CLINICAL TRIAL: NCT04651387
Title: Efficacy and Safety of Ozonised Oil (HOO) as Adjuvant Nutrition Supplement in COVID-19 Patients With Mild-to-Moderate Disease - HOO-COVID Project
Brief Title: Efficacy and Safety of Ozonised Oil (HOO) in COVID-19 Patients
Acronym: HOO-COVID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Patients enrolled
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Licia Iacoviello, Professor, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DEP_052020
Record Dates: First submitted 2020-12-01; First posted 2020-12-03 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV Infection
Keywords: ozone therapy, decrease of viral load of SARS-CoV-2
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In addition to the routine standard treatments for COVID-19, in the intervention group, combined use of "HOO capsules" and "HOO oropharyngeal and nasal spray" will be administered
  Interventions: Dietary Supplement: Ozonized oil (HOO
- Control group (No Intervention): For the control group, the placebo will be not considered and they will follow the routine standard treatments for COVID-19.

INTERVENTIONS:
Dietary Supplement: Ozonized oil (HOO — In addition to the routine standard treatments for COVID-19, in the intervention group, combined use of "HOO capsules" and "HOO oropharyngeal and nasal spray" will be administered 3 times per day (after breakfast, lunch, dinner, possibly with a delay of one hour from the routine treatment) and will be prescribed for 2 weeks (14 days).
  Posology: 3 HOO capsules plus 3 HOO intranasal administrations for each naris plus 3 HOO oropharyngeal administrations.
  Arms: Intervention group

SUMMARY:
The anti-viral efficacy of ozone against RNA viruses is already established. Ozone gas have been already proposed as possible therapy for Covid-19 infection with insofar limited success. The development of ozonized oil (HOO) solved this problems making ozone highly stable and bioavailable due to its bound with the lipid carrier. HOO administration is totally noninvasive occurring by oral administration of pills or as nasal spray.

HOO regimen could be proposed as complimentary therapeutic treatment for Covid-19 infection, without the need of any modifications of the established standard therapeutic protocols. This complimentary treatment, could be helpful to (a) decrease the severity of the diseases lowering the number of Covid-19 patients requiring high-intensity therapies; (b) fasten qPCR negativization after disease and time-span of hospital recovery.

The objective of this study is to investigates the effectiveness of combined use of "HOO capsules" and "HOO oropharyngeal and nasal spray" as a therapeutic supplement in the treatment of patients with confirmed COVID-19, who are moderately ill.

DETAILED DESCRIPTION:
The anti-viral efficacy of ozone against RNA viruses is already established. Ozone gas have been already proposed as possible therapy for Covid-19 infection with insofar limited success. Indeed, in this form, ozone is extremely volatile and its beneficial effects are only transient. Furthermore, in these studies ozone was administered by auto-hemo-transfusion, an invasive approach that cannot be pursued for preventive purposes in healthy subjects or in severely affected patients. The development of ozonized oil (HOO) solved this problems making ozone highly stable and bioavailable due to its bound with the lipid carrier. HOO administration is totally noninvasive occurring by oral administration of pills or as nasal spray.

A challenge test was developed to identify new strategies to prevent Covid-19 infection. Sensitive cells expressing the ACE2 receptor were challenged with oro-pharyngeal containing high viral loads of Covid-19 and the amount of viral RNA able to penetrate inside the cells quantified by qPCR. The ability to inhibit viral infection by UV radiation, hydrogen peroxide, anti-spike Covid-19 antibodies and HOO was comparatively evaluated. The only agent able to fully neutralize Covid-19 was HOO.

The HOO efficacy in preventing finding is due to (a) the high sensitivity of Covid-19 to oxidative stress; (b) the high lipophilicity of Covid-19 and the wide exposure of its lipid envelope for the interaction with lipohilic HOO; (c) the sensitivity of Covid-19 spike proteins to oxidative stress induced by HOO due to their high abundancy of neutrophilic sulphur-rich sites; (d) the HOO capacity to penetrate inside the cells arresting Covid-19 intra-cellular assembly; (e) HOO anti-inflammatory properties causing inhibition of pulmonary macrophage activation, thromboxane release and consequent pulmonary thrombo-embolism, a severe complication occurring in Covid-19 patients; (f) the increased oxygen availability in lung parenchyma.

HOO regimen could be proposed as complimentary therapeutic treatment for Covid-19 infection, without the need of any modifications of the established standard therapeutic protocols. This complimentary treatment, could be helpful to (a) decrease the severity of the diseases lowering the number of Covid-19 patients requiring high-intensity therapies; (b) fasten qPCR negativization after disease and time-span of hospital recovery.

The objective of this study is to investigates the effectiveness of combined use of "HOO capsules" and "HOO oropharyngeal and nasal spray" as a therapeutic supplement in the treatment of patients with confirmed COVID-19, who are moderately ill.

This study is conducted as an open-label, prospective, controlled, multi-center randomized clinical trial on 74 COVID-19 patients (both sex , aged 18-80 years).

In addition to the routine standard treatments for COVID-19, in the intervention group, combined use of "HOO capsules" and "HOO oropharyngeal and nasal spray" will be administered 3 times per day and will be prescribed for 2 weeks (14 days). For the control group, the placebo will be not considered and they will follow the routine standard treatments for COVID-19.

The study is aimed at defining if HOO therapy decreases the viral load of SARS-CoV-2 (main outcome). Additionally, secondary objectives will be the assessment of the temporal profile of viral load, the proportion of patients with virological clearance, the hospitalization duration stay, intensive care admission and time to, the COVID-19 Severity and in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Real time PCR-approved positive COVID-19 test (nasopharyngeal swabs).
* Both gender
* Age between 18 and 80 years
* Lack of participation in other clinical trials
* COVID-19 Severity Score ≤ 5
* Hospitalized ≤48 hours.
* Signing informed consent and willingness of the participant to accept randomization to any assigned treatment

Exclusion Criteria:

* Pregnancy and breastfeeding.
* BMI ≥35 kg/m2
* Severe and critical COVID-19 pneumonia (COVID-19 Severity Score > 5)
* Patient connected to the ventilator
* SaO2 less than 80%
* Having liver failure, chronic hepatitis, cirrhosis, and cholestatic liver diseases
* Any severe medical condition with a prognosis of < 6 months
* Alcohol and drug abuse (during the last 30 days)
* History of known allergy to peanuts

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Viral load of SARS-CoV-2 | up to one week
  The study is aimed at defining if HOO therapy decreases the viral load of SARS-CoV-2 at day 7.

SECONDARY OUTCOMES:
The temporal profile of viral load of SARS-CoV-2 | up to four weeks
  The temporal profile of viral load at baseline, day 7, 14 and 28
The proportion of patients with virological clearance | up to four weeks
  The proportion of patients with virological clearance at day 14 and 28
SaO2 | up to four weeks
  Increasing SaO2, day 7, 14 and 28
hospitalization stay | through study completion, an average of 3 months
  The hospitalization duration stay
Intensive care | through study completion, an average of 3 months
  Intensive care admission and time to
COVID-19 Severity Score | up to four weeks
  The COVID-19 Severity Score at day 14 and 28 Score definition: 1 is "no limitation of activities"; 2 is "limitation of activities"; 3 is "hospitalized, no oxygen therapy"; 4 is " hospitalized, oxygen by mask or nasal prongs"; 5 is "non-invasive ventilation or high-flow oxygen"; 6 is "intubation and mechanical ventilation"; 7 is "ventilation + additional organ support - pressors, RRT (renal replacement therapy), ECMO (extracorporeal membrane oxygenation)", and 8 is "death".
in-hospital mortality | through study completion, an average of 3 months
  Death occurred during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Licia Iacoviello, MD, PhD, Principal Investigator — IRCCS Neuromed

IPD SHARING:
Plan to Share IPD: No